CLINICAL TRIAL: NCT00076362
Title: Pediatric Hypothalamic Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CSMS995B2403
Record Dates: First submitted 2004-01-21; First posted 2004-01-23 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: Sandostatin LAR

SUMMARY:
This trial is being conducted in pediatric patients with Hypothalamic Obesity. This generally occurs in people who have had an injury to or tumor in their hypothalamus (gland or organ that secretes hormones). The purpose of this trial is to see how an investigational treatment controls the hormone insulin by lowering the level of insulin in the body resulting in a weight loss in children who are at least 6 years of age but less than 18 years of age. Some children in this trial will receive placebo.

To qualify for this study, you and your child's doctor must feel that your child's weight is inadequately controlled within a year from the time of injury to the hypothalamus or tumor of the hypothalamus. This study will help to determine if an investigational treatment is of benefit in controlling a child's weight.

ELIGIBILITY:
* Male and female patients ages 6 to less than 18
* Patients who have experienced any form of cranial insult related to cranial trauma, or to a tumor or it's treatment (i.e. surgery, radiation, and/or chemotherapy)
* Patients who are at least one year out following therapy for their tumor
* Patients who have severe cardiovascular dysfunction (for example cardiomyopathy, congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation) will be excluded
* Patients with severe neurologic handicaps which preclude normal physical activity will be excluded.
* Patients confined to bed and those patients who are wheelchair bound which prevents them from activities of daily living or normal physical activity, i.e. walking, will be excluded from the trial
* Your child must be greater than 120% of their ideal body weight for their height or have a body mass index that is greater than or equal to 27.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2004-03; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BMI

SECONDARY OUTCOMES:
Change from baseline in weight, leptin, insulin AUC, C-peptide AUC, amylin AUC, glucose AUC, dietary intake, physical activity, waist-to-hip ratio, visceral and subcutaneous abdominal fat

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (15):
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - Children's Hospital of Orange County, Orange, California
  - University of California at San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Miami Children'S Hopital, Miami, Florida
  - Childrens Memorial Hospital, Chicago, Illinois
  - St. Vincent Children's Center for Cancer and Blood Diseases, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - U of Tennessee HELP Center, Memphis, Tennessee
  - UT Southwestern Children's Medical Center of Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas